CLINICAL TRIAL: NCT02064790
Title: Comparison of Gabapentin and Pregabalin for Cervical and Lumbar Radicular Pain
Brief Title: Comparison of Gabapentin and Pregabalin for Radicular Pain
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Diana Sodiq, Assistant Professor of Orthopaedics, Emory University
Other Study IDs: IRB00069871
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Radicular; Neuropathic, Lumbar, Lumbosacral; Radicular; Neuropathic, Cervical
Keywords: Gabapentin; Pregabalin; Lyrica; Neurontin; lumbar; cervical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group G - receiving gabapentin: Receiving gabapentin as standard of care. No intervention
- Group P - receiving pregabalin: Receiving pregabalin as standard of care No intervention
- Group Z - no neuropathic agent: Receiving only conservative treatment No drug treatment No intervention

SUMMARY:
Although some studies show improvement of pain and associated effects of pain with off-label use of neuropathic agents for cervical or lumbar radiculopathy, there is limited published evidence so far. We propose to complete a year-long prospective, observational study as a pilot to recruit 400 patients within the year and follow their pain level, function, and QOL measures for 16 weeks to determine whether it is feasible to continue studying this group in the future. We expect that pain, function, and quality of life will be improved in the group of patients who are given neuropathic agents as an adjunct to other conservative treatments compared to the expected 65% of patients with similar symptoms who are treated conservatively without neuropathic agents. We do not expect a statistically significant difference between the two neuropathic agents.

Since these drugs are currently used off-label, there is limited empirical evidence regarding which agent is more efficacious compared to the other, and since their use in treating radicular pain is based mostly on anecdotal evidence so far, prescription of one or the other of these agents has been based on likely compliance (medication needed twice a day, three times a day) or whether or not the patients' insurance will pay for one or the other. This study will be a first step to better assist practitioners in counselling their patients on use of these medications in radiculopathy, examining rates of discontinuation due to side effects and what effects these medications have on perceived pain, function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Cervical or lumbar radicular complaints with clinical diagnosis of radiculopathy or sciatica
* Aged 18 years and older
* Able to provide informed consent either with or without a legally authorized representative
* Patients with VAS> or = 4 (Visual Analog Pain score)

Exclusion Criteria:

* Under the age of 18
* Previously completed epidural injections within 3 weeks of the study
* Undergone cervical or lumbar surgery
* History of renal disease, metastatic disease to the spine, vertebral fractures
* Individuals with pending litigation, workers compensation claims or disability claims
* Unable to provide informed consent and no legally authorized representative is available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants of both genders and all ethnicities will be invited to participate in this study as they present to Emory Orthopaedics and Spine Clinic and are diagnosed with and treated for cervical or lumbar radicular pain.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pain reduction with Visual Analogue Scale | 8 weeks
  Specific Aim 1: To determine the efficacy of addition of gabapentin or pregabalin to conservative management for pain reduction in patients with cervical or lumbar radiculopathy.
  Hypothesis 1: There is a significant improvement of pain level with addition of one of the neuropathic agents for patients with radiculopathy compared to patients who are treated without them.

SECONDARY OUTCOMES:
To compare the efficacy of each of the two neuropathic agents to the other in treatment of cervical or lumbar radiculopathy | 8 weeks
  Outcome measures below will be used.
  Oswestry Low Back Pain Disability Questionnaire (ODO) Neck Disability Index (NDI) Usage/Reduction of non-neuropathic pain meds at each interval Side effects of medications

OTHER OUTCOMES:
To determine the rate of compliance and reported side effects related to the neuropathic agent used. | 8 weeks
  Hypothesis:
  There will be a less than 15% discontinuation rate secondary to side effects in either of the two neuropathic agents.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Sodiq, D.O., Principal Investigator — Emory University
Locations (1):
- Emory Orthopaedics and Spine Center, Atlanta, Georgia, United States